CLINICAL TRIAL: NCT03365570
Title: Prevalence of Oral Manifestations of Iron Deficiency Anemia in a Sample of Egyptian Population, Hospital-based Cross-sectional Study
Brief Title: Prevalence of Oral Manifestations of Iron Deficiency Anemia in a Sample of Egyptian Population
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Abdallah Alsheikh, BDS, Master student at oral medicine department, Cairo University
Other Study IDs: oral lesions and anemia
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Iron Deficiency Anemia
Keywords: hemoglobin, iron, oral lesions, oral manifestations,cross-sectional study
MeSH Terms: conditions — Anemia, Iron-Deficiency; Oral Manifestations

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
According to WHO Reportin 2002, iron deficiency anemia was considered to be the most important contributing factor to the global burden of anemia. Children and women in reproductive ages are more at risk factor for developing iron deficiency anemia.No previous study has been held to assess prevalence of oral manifestations of iron deficiency anemia as a hospital-based cross-sectional study on a sample of Egyptian patients in hematology department (no previous data recorded).

DETAILED DESCRIPTION:
Study will be held in at the Hematology department at El Qasr Al-Einy Cairo University Hospital data collection started from February 2018 till end of April 2018 primary completion.

Clinical examination performed for oral mucosa, the number and type of lesions will be recorded. Patients' age, sex, duration of illness, type of anemia, location of any oral lesion or abnormality, history of drug and alcohol consumption, and presence or absence of dentures, will be recorded participants will not followed up and data will be collected prospectively.

A copy of participant's blood record will be obtained from the hematology department upon its approval.

Participants:

Egyptian patients diagnosed with Iron deficiency anemia that attending the Hematology department at El Qasr Al-Einy Cairo University Hospital will be enrolled in the study. The age of participant enroll will be up to 70 years old, males and females will be included.

For each eligible participant, a full history will be obtained according to an assessment sheet, followed by clinical examination which will be done through an interview between the investigator and the patient.

All participants will be asked to sign a study-related informed consent. Oral manifestations of these patients will be evaluated by an oral medicine master student (the investigator).

ELIGIBILITY:
Inclusion Criteria

1. Patients diagnosed with iron deficiency anemia based on their blood tests.
2. Age: by maximum 70 years old.
3. Males and females will be included.

Exclusion Criteria

1. Patients suffering from any other systemic diseases known to influence oral and maxillofacial manifestations will be excluded.
2. Patients suffering from any other systemic diseases known to cause IDA as secondary condition will be excluded.
3. Patients on drug therapy that may have oral mucosal manifestations.
4. Lesions appear because of existing local factors for example traumatic ulcer on the tongue because of sharp tooth against tongue, angular cheilitis because of poor denture design and older age patients.
5. Inflammatory diseases, malignancy, or recent surgery were excluded.

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants:
  Egyptian patients diagnosed with Iron deficiency anemia that attending the Hematology department at El Qasr Al-Einy Cairo University Hospital will be enrolled in the study. The age of participant enroll will be up to 70 years old, males and females will be included.
  For each eligible participant, a full history will be obtained according to an assessment sheet, followed by clinical examination which will be done through an interview between the investigator and the patient.
  All participants will be asked to sign a study-related informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of oral mucosal lesions | 15 minutes
  Presence of oral mucosal lesions will be assessed by clinical picture into dichotomous outcome (Yes/No) and percentage of each.

CONTACTS AND LOCATIONS:
Overall Officials: Fatheya Zahran, Professor, Study Chair — Head of the Department of Oral Medicine and periodontology Cairo University; Eman Alsheikh, Principal Investigator — Master student; Eman Mo Amr, A.Professor, Study Director — associate professor in the Department of Oral Medicine and periodontology Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeLoughery TG. Iron Deficiency Anemia. Med Clin North Am. 2017 Mar;101(2):319-332. doi: 10.1016/j.mcna.2016.09.004. Epub 2016 Dec 8. PMID 28189173
- [Result] Rohani B. Oral manifestations and blood profile in patients with iron deficiency anemia. J Formos Med Assoc. 2015 Jan;114(1):97. doi: 10.1016/j.jfma.2014.07.004. Epub 2014 Aug 10. No abstract available. PMID 25115528
- [Result] Wu YC, Wang YP, Chang JY, Cheng SJ, Chen HM, Sun A. Oral manifestations and blood profile in patients with iron deficiency anemia. J Formos Med Assoc. 2014 Feb;113(2):83-7. doi: 10.1016/j.jfma.2013.11.010. Epub 2013 Dec 30. PMID 24388269